CLINICAL TRIAL: NCT01183273
Title: Prospective Randomized Trial Comparing Laparoscopic Roux-en-y Gastric Bypass to Micro-laparoscopic Roux-en-y Gastric Bypass
Brief Title: Randomized Trial Comparing Laparoscopic Roux-en-y Gastric Bypass to Micro-laparoscopic Roux-en-y Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzanne J. Rose (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor-Investigator, Suzanne J. Rose, Director, Office of Clinical Trials, Danbury Hospital
Organization: Danbury Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29043
Record Dates: First submitted 2010-08-09; First posted 2010-08-17 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micro-laparoscopic bypass (Active Comparator)
  Interventions: Procedure: Microlaparoscopic gastric bypass
- Laparoscopic gastric bypass (Active Comparator)
  Interventions: Procedure: Laparoscopic Surgery

INTERVENTIONS:
Procedure: Microlaparoscopic gastric bypass — microlaparoscopic gastric bypass will be performed using standard of care procedure.
  Arms: Micro-laparoscopic bypass
Procedure: Laparoscopic Surgery — laparoscopic gastric bypass will be performed using standard of care procedure.
  Arms: Laparoscopic gastric bypass

SUMMARY:
Background Laparoscopy is the preferred surgical approach for a number of different diseases as it allows for diagnosis and treatment in the setting of a safe and feasible method offering enhanced cosmesis. The natural evolution of laparoscopy is micro-laparoscopy which utilizes smaller instruments and optics. Technological advancements have enabled miniaturization of the surgical equipment without compromising diagnostic or operative capabilities.

Dr. Keith Zuccala is currently performing micro-laparoscopic gastric bypass with an identical safety profile as traditional laparoscopy (NSQIP data comparison between Dr. Laura Choi and Dr. Keith Zuccala). The current trend in laparoscopy is to minimize incisions and their size to decrease trauma to the abdominal wall.

Study Design Both methods have never been compared in a prospective randomized trial to address the following questions.

1. Is there a difference in outcome?
2. Is there a decrease in postoperative pain?
3. Does it decrease time off from work?
4. Does micro-laparoscopy increase OR time?
5. What is the effect on cost of micro-laparoscopy? Patients will be randomized to one or the other method, disclosing that to the investigators best knowledge both methods are equally safe and that Dr. Zuccala has performed several hundred cases using both methods.

Patient Population Projected sample size would be 50 patients in each group. Accrual should be feasible over the course of 9-12 months.

Data collection (patients will be followed for a total of 30 days for the purpose of this study)

1. NSQIP data to assess outcome
2. Postoperative usage of pain medication while in the hospital
3. Time off from work
4. OR time
5. Direct cost of procedure as it relates to material used

DETAILED DESCRIPTION:
This study compares two groups of patients who have voluntarily chosen to undergo roux-n-y gastric bypass surgery. The groups will be randomized to receive micro-laparoscopic or laparoscopic surgery to be performed by the same surgeon, Dr. Keith Zuccala.

Study Schema

* The patient attends an informational seminar conducted by the Bariatric Surgery Department
* The patient is scheduled for an initial consultation with the bariatric PA/NP where the patient provides: a letter of referral for Bariatric Surgery from primary care doctor or specialty physician; insurance referral; and assurance that health insurance coverage includes Bariatric Surgery.
* Following the initial consultation, the patient is scheduled for the following: comprehensive blood testing; psychological screening/evaluation; dietary evaluation; appointment with the surgeon; pulmonary evaluation (if needed); cardiology evaluation (if needed); gastroenterology evaluation (if needed).
* An appointment for medical clearance with the referring surgeon is scheduled and completed within three weeks of surgery. At this appointment an electrocardiogram (EKG) and repeat blood work will be carried out.
* The patient is deemed to meet all inclusion criteria.
* The patient is advised to follow all pre-operative instructions as advised by the nursing staff and explained in the Danbury Hospital Center for Weight Loss Surgery Guide.
* Surgical procedures performed are standard for those already utilized daily in the surgery department for gastric bypass procedures.
* The patient is closely observed in the hospital and given specific discharge instructions upon leaving the hospital
* The patient is followed for a maximum of 60 days after surgery and asked how many days of work they missed.
* The NSQIP data base and patient medical record are used to assess outcome, postoperative pain, OR time and surgery cost

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI) ≥ 40 with or without co-morbid conditions*
* A BMI ≥ 35 with co-morbid conditions*
* Permanent lifestyle changes including exercise
* No significant, untreated psychiatric illnesses
* Age ≥ 18 years
* Sufficient ability and cognition to understand surgery, potential complications and subsequent associated changes
* Willingness to participate in treatment and long-term follow-up
* Proof of failed attempts at non-surgical weight reduction
* Acceptable medical/operative risks * Co-morbid solutions include: hypertension, diabetes mellitus, cardiac disease, hypercholesterolemia/hyperlipidemia, sleep apnea, asthma, hypoventilation syndrome of obesity, degenerative joint disease, gastro-esophageal reflux disease, venous stasis ulcers, depression, menstrual irregularities/infertility, polycystic ovary syndrome, fungal skin infections.

Exclusion Criteria:

* The need to convert from laparoscopic roux-n-y to an open abdominal procedure.
* Patients with congestive heart failure or other serious illness which would prevent the patient from a successful surgery and recovery
* Women who are nursing or pregnant
* Patients who smoke
* Patient's insurance will not cover the cost of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety of micro-laparoscopic versus laparoscopic gastric bypass | 2 years

SECONDARY OUTCOMES:
Postoperative pain | 30 days
Time off from work | 30 days
Operating Cost | The time of surgery is collected following patient discharge approximately 4 to 5 days
Time of Surgery | The time of surgery is collected following patient discharge approximately 4 to 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Saldinger, M.D., Study Chair — Danbury Hospital; Keith Saldinger, M.D., Principal Investigator — Danbury Hospital; Suzanne J House, M.S., Ph.D., Study Director — Danbury Hospital
Locations (1):
- Danbury Hospital, Danbury, Connecticut, United States